CLINICAL TRIAL: NCT07014228
Title: Evaluation of Post Operative Pain in Non-surgical Endodontic Retreatment in Single vs Multiple Visits
Brief Title: Evaluation of Post-operative Pain During Retreatment in Different Visits
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Armed Forces Institute of Dentistry, Pakistan (Other)
Responsible Party: Principal Investigator, Ahmed Abdullah, Principal investigator, Armed Forces Institute of Dentistry, Pakistan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Re-endo pain comparison
Record Dates: First submitted 2025-06-01; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Patients will be divided into two equal groups and given two different interventions (single vs. multi-visit reendo).
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single visit group (Experimental): Endodontic retreatment in this group will be performed in a single visit. Initiated, deobturated, disinfection done and completed during the same visit.
  Interventions: Procedure: single visit re-endo
- Multi visit Group (Active Comparator): Endodontic retreatment in this group will be performed in more than 1 visit. The retreatment will be initiated, deobturated, and disinfection done and completed in second or third visits..
  Interventions: Procedure: multi visit re-endo

INTERVENTIONS:
Procedure: single visit re-endo — In this group, a single visit re-endodontic treatment will be performed and completed in the same visit, including all the steps.
  Arms: Single visit group
Procedure: multi visit re-endo — In this group, a multi-visit re-endodontic treatment will be performed and completed over different visits, including all the steps.
  Arms: Multi visit Group

SUMMARY:
Endodontic retreatment is performed to alleviate symptoms of recurring infection, post-treatment disease after primary endodontic therapy. Retreatment can be performed in either single or multiple visits. and have their own implications. it is important to compare the patient response and post-op pain after single vs multi-visit reendo treatment.

DETAILED DESCRIPTION:
Introduction:

Treating endodontic failure cases has always been a challenge for the clinician due to the complex nature of disease which includes resistant microorganisms, iatrogenic errors and cleaning and shaping of un-instrumented areas. Endodontic retreatment can be done in either single or multiple visits. Multiple visits have the added advantage of placement of intracanal medicament resulting in decreased bacterial load and reduced pain, whereas single visit endodontic retreatment reduces chances of inter appointment microbial contamination. This study aims to evaluate post operative pain among both groups.

Objective:

To evaluate frequency of post-operative pain in endodontic retreatment cases after single vs multiple (two) visits root canal therapy.

Materials and Methods:

STUDY SETTING: Department of Operative Dentistry, AFID Rawalpindi.

ELIGIBILITY:
Inclusion Criteria:

* Patients with unremarkable/ noncontributory medical history
* Age range between 15-45 years
* Cases of failed endodontic treatment resulting from inadequate root filling
* No systemic disease
* No periodontal disease

Exclusion Criteria:

* Patients having teeth with periodontal pathology
* root fractures
* Immature root apices
* Endodontic posts
* Root perforations
* Immunocompromised health were excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Post operative pain after re-endo | 6 hours - 72 hours
  Post-operative pain after single vs multi visit re-endo treatment to be compared. The patients will be guided in detail about the procedure and how to document their response to the treatment. The Visual Analog Scale (VAS). numbered from 0-10, with 0 being no pain, 1 - 3: mild pain, 4-6: moderate pain, and 7-10 severe pain, will be used to record pain experienced by the patients and notified to the investigator.

CONTACTS AND LOCATIONS:
Locations (1):
- Armed Forces Institute of dentistry, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No